CLINICAL TRIAL: NCT04009577
Title: A Multicenter, Pilot Study to Evaluate Next-Dose Transition From Zolpidem to Lemborexant for the Treatment of Insomnia
Brief Title: A Study to Evaluate Next-Dose Transition From Zolpidem to Lemborexant (LEM) for the Treatment of Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2006-A001-312
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2020-02

CONDITIONS: Insomnia
Keywords: Insomnia; Sleep Initiation and Maintenance Disorders; Insomnia Disorder; Sleeplessness; E2006; Zolpidem; Lemborexant
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — leukocyte endogenous mediator; lemborexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (LEM 5 mg) (Experimental): Participants who were taking zolpidem tartrate (ZOL) at least 3 but fewer than 5 nights per week, for each of at least 2 weeks of the 3-week Screening Period, will initially receive LEM 5 mg administered as a tablet, orally for up to 2 weeks.
  Participants who meet both criteria for intermittent (Cohort 1) and frequent ZOL use (Cohort 2A and 2B) for 1 week each of the last 2 weeks of the 3-week Screening Period will be assigned to Cohort 1 and also will receive LEM 5mg.
  Interventions: Drug: LEM 5 mg
- Cohort 2A (LEM 5 mg) (Experimental): Participants who were taking ZOL at least 5 nights per week, during, at minimum, the last 2 weeks of the 3-week Screening Period, will initially receive LEM 5 mg administered as a tablet, orally for up to 2 weeks.
  Interventions: Drug: LEM 5 mg
- Cohort 2B (LEM 10 mg) (Experimental): Participants who were taking ZOL at least 5 nights per week, during, at minimum, the last 2 weeks of the 3-week Screening Period, will initially receive LEM 10 mg administered as a tablet, orally for up to 2 weeks.
  Interventions: Drug: LEM 10 mg

INTERVENTIONS:
Drug: LEM 5 mg — LEM tablet.
  Other Names: E2006; Lemborexant
  Arms: Cohort 1 (LEM 5 mg); Cohort 2A (LEM 5 mg)
Drug: LEM 10 mg — LEM tablet.
  Other Names: E2006; Lemborexant
  Arms: Cohort 2B (LEM 10 mg)

SUMMARY:
The primary objective of the study is to evaluate the proportion of adult [greater than or equal to (>=) 18 years] participants with insomnia disorder taking zolpidem tartrate immediate release (ZOL-IR) or zolpidem tartrate extended release (ZOL-ER), intermittently or frequently, who transition to lemborexant 5 milligram (mg) (LEM5) or 10 mg (LEM10) after 2 weeks of receiving LEM.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the Diagnostic and Statistical Manual of Mental Disorders, 5th ed (DSM-5) criteria for Insomnia Disorder, either currently or prior to zolpidem use, as follows:

   * Complains of dissatisfaction with nighttime sleep, in the form of difficulty staying asleep and/or awakening earlier in the morning than desired despite adequate opportunity for sleep
   * Frequency of complaint >=3 times per week
   * Duration of complaint >=3 months
   * Associated with complaint of daytime impairment
2. Reports spending at least 7 hours in bed per night
3. History of intermittent [taking zolpidem at least 3 or 4 nights per week], or frequent use (at least 5 nights per week) of ZOL-IR or ZOL-ER, for at least 1 month
4. Confirmation of intermittent or frequent use of zolpidem (based on review of drug use data). Intermittent use is defined as taking zolpidem at least 3 but fewer than 5 nights per week, for at least 2 weeks each of the 3-week Screening Period. Frequent use is defined as taking zolpidem at least 5 nights per week, during, at minimum, the last 2 weeks of the 3-week Screening Period
5. Willing and able to comply with all aspects of the protocol, including staying in bed for at least 7 hours each night
6. Willing not to start another pharmacologic treatment for the management of insomnia during the participant's participation in the study

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at screening or baseline (as documented by a positive serum pregnancy test). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
2. Females of childbearing potential who:

   Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:
   * total abstinence (if it is their preferred and usual lifestyle)
   * an intrauterine device or intrauterine hormone-releasing system (IUS)
   * a contraceptive implant
   * an oral contraceptive (Participant must be on a stable dose of the same oral contraceptive product for at least 28 days before dosing and throughout the study and for 28 days after study drug discontinuation)
   * have a vasectomized partner with confirmed azoospermia
   * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)
3. Any history of moderate or severe obstructive sleep apnea (OSA)
4. Current evidence of a clinically significant, active respiratory disorder other than mild OSA. This includes bronchiectasis, emphysema, asthma, chronic obstructive pulmonary disease or any other pulmonary disorder identified by review of medical history or physical examination, and which in the opinion of the investigator, could compromise the participant's safety or interfere with study assessments
5. A current diagnosis of periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, or an exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia as follows:

   * STOP-Bang score >=5 (participants previously diagnosed with mild OSA are not excluded)
   * International Restless Legs Scale (IRLS) score >=16
6. Habitually naps during the day more than 3 times per week
7. Reports symptoms potentially related to narcolepsy, that in the clinical opinion of the investigator indicates the need for referral for a diagnostic evaluation for the presence of narcolepsy
8. Reports a history of sleep-related violent behavior, or sleep driving, or any other complex sleep-related behavior (eg, making phone calls or preparing and eating food while sleeping), whether spontaneous or associated with a pharmacological sleep agent
9. Takes a dose of ZOL-IR greater (>)10 mg per night, or ZOL-ER >12.5 mg per night
10. Takes a dose of zolpidem that is lower than what is prescribed
11. Reports having altered zolpidem tablets
12. Unwilling to forgo alcohol consumption within 3 hours of bedtime for the duration of participation in the study
13. Used any prohibited prescription or over-the-counter concomitant medications within 1-week or 5 half-lives, whichever is longer, before the first dose of study medication (A list of prohibited concomitant medications is presented in the protocol)
14. Used any pharmacologic modality of treatment for insomnia other than zolpidem, including marijuana, within 1-week or 5 half-lives, whichever is longer, before the Screening Period
15. A prolonged difference between QTc corrected by Fridericia's formulas (QTcF) interval [QTcF >450 millisecond (ms)] as demonstrated by a repeated electrocardiogram
16. Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening (ie, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale [C-SSRS])
17. Any lifetime suicidal behavior (per the Suicidal Behavior section of the C-SSRS)
18. Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, and renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments. Participants for whom a sedating drug would be contraindicated for safety reasons because of the participant's occupation or activities are also excluded
19. Hypersensitivity to LEM or any of the excipients
20. Any history of or concomitant medical condition that in the opinion of the investigator(s) would compromise the participant's ability to safely complete the study
21. Planned surgery that requires general, spinal, or epidural anesthesia that would take place during the study. Planned surgery, which requires only local anesthesia and which can be undertaken as a day case without inpatient stay postoperatively, need not result in exclusion if in the opinion of the investigator this operation does not interfere with the study procedures and patient safety
22. Psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics or prior suicide attempt(s) within approximately the last 2 years
23. History of drug or alcohol dependency or abuse within approximately the last 2 years
24. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5 times the half-life, whichever is longer, preceding informed consent
25. Previously participated in any clinical trial of LEM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - PACT, Glendale, Arizona
  - Northern California Research Corp, Sacramento, California
  - Artemis Institute For Clinical Research LLC - San Diego - ClinEdge - PPDS, San Diego, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Fleming Island Center For Clinical Research - ERN-PPDS, Fleming Island, Florida
  - MD Clinical, Hallandale, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - NeuroTrials Research Inc. - BTC - PPDS, Atlanta, Georgia
  - SleepCare Research Institute Inc, Stockbridge, Georgia
  - Chicago Research Center Inc - ClinEdge - PPDS, Chicago, Illinois
  - Centennial Medical Group - Elkridge - Rx Trials, Elkridge, Maryland
  - Albuquerque Neurosciences Inc, Albuquerque, New Mexico
  - Clinilabs Drug Development Corporation, New York, New York
  - CTI Clinical Research Center - ClinEdge - PPDS, Cincinnati, Ohio
  - Clinical Neuroscience Solutions Inc, Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website https://eisaiclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 17 investigative sites in the United States from 15 July 2019 to 26 June 2020. This study included 2 parts: Core study (Pretreatment phase and Treatment Phase) and Extension Phase.
Pre-assignment Details: A total of 99 participants were screened, of which 46 were screen failures and 53 participants were enrolled and randomized into the Core study. Out of 53 randomized and treated participants in the Core Study, 43 participants entered Extension Phase and 41 participants received study drug.
Groups:
- Cohort 1A: LEM 5 or LEM 10 (Intermittent ZOL Use): Participants who took zolpidem tartrate (ZOL) at least 3 nights but fewer than 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received lemborexant 5 milligram (mg) (LEM5) or 10 mg (LEM10) tablet up titrated (in case previous dose was ineffective), orally, once at night for up to 2 weeks in Titration Period of Core Study and continued to receive LEM5 or LEM10 tablet up titrated (in case previous dose was ineffective), orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 1B: LEM 5 or LEM 10 (Mixed ZOL Use): Participants who met both criteria for intermittent and frequent ZOL use for 1 week each of the last 2 weeks of the 3-week Screening Period, initially received LEM5 or LEM10 tablet up titrated (in case previous dose was ineffective), orally, once at night for up to 2 weeks in Titration Period of Core Study and continued to receive LEM5 or LEM10 tablet up titrated (in case previous dose was ineffective), orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 2A: LEM 5 or LEM 10 (Frequent ZOL Use): Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM5 or LEM10 tablet up titrated (in case previous dose was ineffective), orally, once at night for up to 2 weeks in Titration Period of Core Study and continued to receive LEM5 or LEM10 tablet up titrated (in case previous dose was ineffective), orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 2B: LEM 10 or LEM 5 (Frequent ZOL Use): Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM10 or LEM5 tablet down titrated (due to tolerability), orally, once at night for up to 2 weeks in Titration Period of Core Study and continued to receive LEM10 or LEM5 tablet down titrated (due to tolerability), orally, once at night for up to 12 weeks in the Extension Phase.
Period: Core Study
Arm/Group | Cohort 1A: LEM 5 or LEM 10 (Intermittent ZOL Use) | Cohort 1B: LEM 5 or LEM 10 (Mixed ZOL Use) | Cohort 2A: LEM 5 or LEM 10 (Frequent ZOL Use) | Cohort 2B: LEM 10 or LEM 5 (Frequent ZOL Use)
Started | 7 | 3 | 21 | 22
LEM5 | 7 | 3 | 21 | 5
LEM10 | 3 | 2 | 10 | 22
Completed | 6 | 3 | 17 | 17
Not Completed | 1 | 0 | 4 | 5
Not completed — Adverse Event | 1 | 0 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 1
Period: Extension Phase
Arm/Group | Cohort 1A: LEM 5 or LEM 10 (Intermittent ZOL Use) | Cohort 1B: LEM 5 or LEM 10 (Mixed ZOL Use) | Cohort 2A: LEM 5 or LEM 10 (Frequent ZOL Use) | Cohort 2B: LEM 10 or LEM 5 (Frequent ZOL Use)
Started (Participants who completed the Core Study had the option to participate in the Extension Phase) | 6 | 3 | 17 | 17
Treated | 6 | 3 | 15 | 17
LEM5 | 6 | 3 | 15 | 8
LEM10 | 5 | 3 | 12 | 17
Completed | 6 | 3 | 13 | 16
Not Completed | 0 | 0 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Inadequate therapeutic effect | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Not Treated | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included participants who received at least 1 dose of lemborexant.
Groups:
- Cohort 1A: LEM 5 or LEM 10 (Intermittent ZOL Use): Participants who took ZOL at least 3 nights but fewer than 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM5 or LEM10 tablet up titrated (in case previous dose was ineffective), orally, once at night for up to 2 weeks in Titration Period of Core Study and continued to receive LEM5 or LEM10 tablet up titrated (in case previous dose was ineffective), orally, once at night for up to 12 weeks in the Extension Phase.
- Total: Total of all reporting groups
Arm/Group | Cohort 1A: LEM 5 or LEM 10 (Intermittent ZOL Use) | Cohort 1B: LEM 5 or LEM 10 (Mixed ZOL Use) | Cohort 2A: LEM 5 or LEM 10 (Frequent ZOL Use) | Cohort 2B: LEM 10 or LEM 5 (Frequent ZOL Use) | Total
Number analyzed (Participants) | 7 | 3 | 21 | 22 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (6.12) | 60.0 (8.72) | 52.7 (13.57) | 63.5 (10.44) | 59.0 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 14 | 14 | 35
  Male | 3 | 0 | 7 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 6 | 5 | 13
  Not Hispanic or Latino | 6 | 2 | 15 | 17 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 5 | 3 | 10
  White | 6 | 2 | 15 | 18 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Overall Participants Who Transitioned to LEM at the End of the Titration Period of Core Study
Description: Transition to LEM was defined as participant who remained on LEM at the end of the 2-week titration period and either 1) entered the extension phase, or 2) chooses to not enter the extension phase for reasons not related to LEM (including, but not limited to, time commitment related to the study, study-related travel expenses or preference to continue insomnia management with another health care provider).
Time Frame: Up to 2 Weeks
Population: The FAS included participants who received at least 1 dose of lemborexant.
Measure: Number; unit: percentage of participants
Groups:
- Overall Cohort: Participants who took ZOL at least 3 but fewer than 5 nights per week, for the last 2 weeks of the 3-week Screening Period or who met both criteria for intermittent and frequent ZOL use for 1 week each of the last 2 weeks of the 3-week Screening or who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, received LEM5 or LEM10 tablet (as per titration schedule), orally once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed 2 weeks in Titration Period of Core Study continued to receive LEM5 or LEM10 (as per titration schedule) tablet, orally, once at night for up to 12 weeks in the Extension Phase.
Arm/Group | Overall Cohort
Number analyzed (Participants) | 53
percentage of participants | 81.1

2. Secondary Outcome: Percentage of Participants Who Transitioned to LEM at the End of the 2-Week Titration Period of Core Study Within Each Cohort
Description: as for outcome 1
Time Frame: Up to 2 Weeks
Population: The FAS included participants who received at least 1 dose of lemborexant.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1A: LEM 5 or LEM 10 (Intermittent ZOL Use) | Cohort 1B: LEM 5 or LEM 10 (Mixed ZOL Use) | Cohort 2A: LEM 5 or LEM 10 (Frequent ZOL Use) | Cohort 2B: LEM 10 or LEM 5 (Frequent ZOL Use)
Number analyzed (Participants) | 7 | 3 | 21 | 22
percentage of participants | 85.7 | 100 | 81.0 | 77.3

3. Secondary Outcome: Percentage of Participants in the LEM5 Treatment Groups With Dose Increasing to LEM10 at the End of the Titration Period of Core Study by Cohort and Overall
Description: This outcome measure was planned for Cohort 1A, 1B and 2A. As there was no dose increase happened in Cohort 2B, this Outcome Measure is not applicable for Cohort 2B.
Time Frame: Up to 2 Weeks
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: percentage of participant
Arm/Group | Cohort 1A: LEM 5 or LEM 10 (Intermittent ZOL Use) | Cohort 1B: LEM 5 or LEM 10 (Mixed ZOL Use) | Cohort 2A: LEM 5 or LEM 10 (Frequent ZOL Use) | Overall Cohort
Number analyzed (Participants) | 7 | 3 | 21 | 31
percentage of participant | 42.9 | 66.7 | 47.6 | 48.4

4. Secondary Outcome: Percentage of Participants in LEM10 Treatment Group With Dose Decreasing to LEM5 at the End of the Titration Period of Core Study in Cohort 2
Description: This outcome measure was planned for Cohort 2B. As dose decrease happened in Cohort 2B only, this Outcome Measure is not applicable for Cohort 1A, 1B and 2A.
Time Frame: Up to 2 Weeks
Population: The FAS included participants who received at least 1 dose of lemborexant.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2B: LEM 10 or LEM 5 (Frequent ZOL Use)
Number analyzed (Participants) | 22
percentage of participants | 22.7

5. Secondary Outcome: Percentage of Participants With Positive Medication Effect Rating on Each Patient Global Impression of Insomnia (PGI-I) Item at the End of the 2-Week Titration Period of Core Study by Cohort and Overall Using End of the Titration Period Treatment
Description: The PGI-I was a self-report assessment of participant perception of the effects of a medication on their sleep. The PGI-I had 3 items related to study medication effects (a) helped/worsened sleep, (b) decreased/increased time to fall asleep, (c) increased/decreased total sleep time, and 1 item related to perceived appropriateness of study medication strength. The first 3 items were answered on a 3-point scale (1=positive medication effect, 2=neutral medication effect, 3=negative medication effect) and the last item on a different 3 point scale (medication: 1=too strong, 2=just right, 3=too weak), only 'positive medication effects' and 'just right' are reported here.
Time Frame: Up to 2 Weeks
Population: The FAS included participants who received at least 1 dose of lemborexant.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1A: LEM 5 or LEM 10 (Intermittent ZOL Use) | Cohort 1B: LEM 5 or LEM 10 (Mixed ZOL Use) | Cohort 2A: LEM 5 or LEM 10 (Frequent ZOL Use) | Cohort 2B: LEM 10 or LEM 5 (Frequent ZOL Use) | Overall Cohort
Number analyzed (Participants) | 7 | 3 | 21 | 22 | 53
percentage of participants
  Positive medication effect: on Sleep | 42.9 | 66.7 | 33.3 | 54.5 | 43.4
  Positive medication effect: Time to fall asleep | 85.7 | 66.7 | 47.6 | 54.5 | 50.9
  Positive medication effect: Total sleep time | 42.9 | 66.7 | 28.6 | 45.5 | 39.6
  Appropriateness of Medication Strength: Just Right | 71.4 | 100 | 38.1 | 50.0 | 54.7

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 22 weeks
Groups:
- Cohort 1A (Core Study): LEM 5: Participants who took ZOL at least 3 but fewer than 5 nights per week, for the last 2 weeks of the 3-week Screening Period, received LEM5 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study.
- Cohort 1A (Core Study): LEM 10: Participants who took ZOL at least 3 but fewer than 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM5 and later up titrated to LEM10 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study.
- Cohort 1B (Core Study): LEM 5: Participants who met both criteria for intermittent and frequent ZOL use for 1 week each of the last 2 weeks of the 3-week Screening Period, received LEM5 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study.
- Cohort 1B (Core Study): LEM 10: Participants who met both criteria for intermittent and frequent ZOL use for 1 week each of the last 2 weeks of the 3-week Screening Period, initially received LEM5 and later up titrated to LEM10 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study.
- Cohort 2A (Core Study): LEM 5: Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, received LEM5 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study.
- Cohort 2A (Core Study): LEM 10: Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM5 and later up titrated to LEM10 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study.
- Cohort 2B (Core Study) : LEM 5: Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM10 and later down titrated to LEM5 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study.
- Cohort 2B (Core Study): LEM 10: Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, received LEM10 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study.
- Cohort 1A (Extension Phase): LEM 5: Participants who took ZOL at least 3 but fewer than 5 nights per week, for the last 2 weeks of the 3-week Screening Period, received LEM5 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed Titration Period of Core Study entered Extension Phase and continued to receive LEM5 tablet, orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 1A (Extension Phase): LEM 10: Participants who took ZOL at least 3 but fewer than 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM5 and later up titrated to LEM10 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed Titration Period of Core Study entered Extension Phase and continued to receive LEM10 tablet, orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 1B (Extension Phase): LEM 5: Participants who met both criteria for intermittent and frequent ZOL use for 1 week each of the last 2 weeks of the 3-week Screening Period, received LEM5 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed Titration Period of Core Study entered Extension Phase and continued to receive LEM5 tablet, orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 1B (Extension Phase): LEM 10: Participants who met both criteria for intermittent and frequent ZOL use for 1 week each of the last 2 weeks of the 3-week Screening Period, initially received LEM5 and later up titrated to LEM10 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed Titration Period of Core Study entered Extension Phase and continued to receive LEM10 tablet, orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 2A (Extension Phase): LEM 5: Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, received LEM5 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed Titration Period of Core Study entered Extension Phase and continued to receive LEM5 tablet, orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 2A (Extension Phase): LEM 10: Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM5 and later up titrated to LEM10 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed Titration Period of Core Study entered Extension Phase and continued to receive LEM10 tablet, orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 2B (Extension Phase): LEM 5: Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, initially received LEM10 and later down titrated to LEM5 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed Titration Period of Core Study entered Extension Phase and continued to receive initially LEM10 and later down titrated to LEM5 tablet, orally, once at night for up to 12 weeks in the Extension Phase.
- Cohort 2B (Extension Phase): LEM 10: Participants who took ZOL at least 5 nights per week, for the last 2 weeks of the 3-week Screening Period, received LEM10 tablet, orally, once at night for up to 2 weeks in Titration Period of Core Study. Eligible participants who completed Titration Period of Core Study entered Extension Phase and continued to receive LEM10 tablet, orally, once at night for up to 12 weeks in the Extension Phase.
Arm/Group | Cohort 1A (Core Study): LEM 5 | Cohort 1A (Core Study): LEM 10 | Cohort 1B (Core Study): LEM 5 | Cohort 1B (Core Study): LEM 10 | Cohort 2A (Core Study): LEM 5 | Cohort 2A (Core Study): LEM 10 | Cohort 2B (Core Study) : LEM 5 | Cohort 2B (Core Study): LEM 10 | Cohort 1A (Extension Phase): LEM 5 | Cohort 1A (Extension Phase): LEM 10 | Cohort 1B (Extension Phase): LEM 5 | Cohort 1B (Extension Phase): LEM 10 | Cohort 2A (Extension Phase): LEM 5 | Cohort 2A (Extension Phase): LEM 10 | Cohort 2B (Extension Phase): LEM 5 | Cohort 2B (Extension Phase): LEM 10
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/3 | 0/2 | 0/21 | 0/10 | 0/5 | 0/22 | 0/6 | 0/5 | 0/3 | 0/3 | 0/15 | 0/12 | 0/8 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 0/3 | 0/2 | 0/21 | 0/10 | 0/5 | 0/22 | 0/6 | 0/5 | 0/3 | 0/3 | 0/15 | 0/12 | 0/8 | 1/17
Other Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 0/3 | 0/2 | 2/21 | 0/10 | 0/5 | 6/22 | 0/6 | 0/5 | 0/3 | 0/3 | 0/15 | 0/12 | 0/8 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A (Core Study): LEM 5 (N=7) | Cohort 1A (Core Study): LEM 10 (N=3) | Cohort 1B (Core Study): LEM 5 (N=3) | Cohort 1B (Core Study): LEM 10 (N=2) | Cohort 2A (Core Study): LEM 5 (N=21) | Cohort 2A (Core Study): LEM 10 (N=10) | Cohort 2B (Core Study) : LEM 5 (N=5) | Cohort 2B (Core Study): LEM 10 (N=22) | Cohort 1A (Extension Phase): LEM 5 (N=6) | Cohort 1A (Extension Phase): LEM 10 (N=5) | Cohort 1B (Extension Phase): LEM 5 (N=3) | Cohort 1B (Extension Phase): LEM 10 (N=3) | Cohort 2A (Extension Phase): LEM 5 (N=15) | Cohort 2A (Extension Phase): LEM 10 (N=12) | Cohort 2B (Extension Phase): LEM 5 (N=8) | Cohort 2B (Extension Phase): LEM 10 (N=17)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A (Core Study): LEM 5 (N=7) | Cohort 1A (Core Study): LEM 10 (N=3) | Cohort 1B (Core Study): LEM 5 (N=3) | Cohort 1B (Core Study): LEM 10 (N=2) | Cohort 2A (Core Study): LEM 5 (N=21) | Cohort 2A (Core Study): LEM 10 (N=10) | Cohort 2B (Core Study) : LEM 5 (N=5) | Cohort 2B (Core Study): LEM 10 (N=22) | Cohort 1A (Extension Phase): LEM 5 (N=6) | Cohort 1A (Extension Phase): LEM 10 (N=5) | Cohort 1B (Extension Phase): LEM 5 (N=3) | Cohort 1B (Extension Phase): LEM 10 (N=3) | Cohort 2A (Extension Phase): LEM 5 (N=15) | Cohort 2A (Extension Phase): LEM 10 (N=12) | Cohort 2B (Extension Phase): LEM 5 (N=8) | Cohort 2B (Extension Phase): LEM 10 (N=17)
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT04009577/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT04009577/SAP_001.pdf